CLINICAL TRIAL: NCT03329144
Title: Building Resilience in Young Mothers: A CBT-Based Curriculum
Brief Title: CBT for Young Mothers
Acronym: CBTYM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Strive Niagara (Unknown); Niagara Region Public Health (Other)
Responsible Party: Principal Investigator, Ryan Van Lieshout, MD, PhD, Assistant Professor, Department of Psychiatry and Behavioural Neurosciences, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBT YM
Record Dates: First submitted 2017-10-30; First posted 2017-11-01 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Anxiety; Depression; Emotion Regulation
Keywords: Young mother; Depression; Anxiety; Resilience; Emotion regulation; Parenting; CBT
MeSH Terms: conditions — Anxiety Disorders; Depression; Emotional Regulation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioural Therapy (Experimental): The women in this arm will receive a 9-week CBT-based curriculum delivered by Public Health Nurses to help build resilience and optimize mood, anxiety, and emotion regulation while attending a supported school program in Niagara Region.
  Interventions: Behavioral: Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — The transdiagnostic CBT-based curriculum is based on the extensive clinical experience of the research team with young women and those struggling with perinatal mental disorders. The team also has significant expertise delivering CBT for depression and anxiety (including perinatal variants) in groups. The manual was developed by the research team and is based on the state-of-the-art in resilience and CBT interventions in adolescents and young adults (e.g., the Penn Resiliency Program (60), Treatment for Adolescent Depression Study (61)). After it was developed, it was subjected to further scrutiny by public health nurses and STRIVE staff, who have extensive experience working with young mothers.

SUMMARY:
Approximately 1 in 4 adolescent mothers will develop depression after delivering a child, though some studies suggest that as many as 53% will develop postpartum depression. A frequent accompanying symptom is emotion dysregulation which not only adversely affects their mental well-being, but jeopardizes their parenting and their child's health. Unfortunately significant barriers exist for young mothers, preventing access to treatment. This study will pilot the feasibility of having public health nurses deliver this 9-session program within a curriculum for teen mothers.

DETAILED DESCRIPTION:
Up to 50% of women who become parents during the teenage years suffer from mental disorders after the birth of their children. While they most commonly develop depression, anxiety problems and substance use disorders are also common, and in many cases they are comorbid. A significant proportion of these young women will also manifest impairing but sub-syndromal levels of symptoms. A frequent accompanying symptom is emotion dysregulation which not only adversely affects their mental well-being, but jeopardizes their parenting and their child's health, as well as longer-term labour market outcomes.

Perinatal mental disorders are associated with significant suffering and high health care costs. Indeed, a single case of postpartum depression is estimated to cost $150,000, a figure that may be even higher in young mothers. Compounding these adverse effects is the fact that just 15% of women with young children and mental disorders receive evidence-based care, numbers that are almost certainly lower in young mothers given their well-known difficulties engaging in health care.

Getting these young women to engage in treatment can be a significant challenge, but given the substantial risks and costs associated with mental disorders in this group, as well as the effectiveness of preventive and treatment interventions (particularly the psychotherapies), it is important that innovative ways to engage and support adolescent mothers be developed. Since many will attend school either in a traditional or adapted setting, the educational system provides an ideal place to deliver interventions aimed at optimizing the mental health of teenage mothers.

The purpose of this pilot study is to develop and establish the feasibility of having public health nurses deliver a 9-session group cognitive behavioural therapy-based resilience curriculum within a school program for teenage mothers at the District School Board of Niagara. In addition to establishing the feasibility and acceptability of the curriculum, estimates of intervention effect and its variance will be generated to support a later large-scale study aimed at assessing its effectiveness.

CBT-based curriculum has been developed to help build resilience and optimize mood, anxiety, and emotion regulation in 15-24 year old women attending a supported school program in Niagara Region. Sixty women will be recruited and changes in depression, anxiety, emotion regulation, parenting, and behavioural problems in their children will be measured pre-group, immediately post-group, and 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* As this is a study of young mothers, women who are 15-24 years of age, speak English, and have a child under the age of 5 will be recruited.

Exclusion Criteria:

* Only women aged 15-24 years who have a child under the age of five will be eligible. Women must be enrolled in the Strive Niagara program.

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of delivering the group | 12 months
  The feasibility of delivering the group will be assessed using simple counts of the number of women who agree to participate

SECONDARY OUTCOMES:
The Beck Depression Inventory | 6 months
  The Beck Depression Inventory is a 21-item scale that assesses the emotional, cognitive, and somatic symptoms of depression.
The Beck Anxiety Inventory | 6 months
  The Beck Anxiety Inventory is a 21-item self-report scale that taps generalized anxiety disorder, the most common comorbidity of depression.
Difficulties in Emotion Regulation Scale | 6 months
  The Difficulties in Emotion Regulation Scale is a 36-item measure of this construct validated in adolescents.
Adult-Adolescent Parenting Inventory | 6 months
  The Adult-Adolescent Parenting Inventory-2 is a validated 40-item measure used to assess strengths and weaknesses in child rearing.
Strengths and Difficulties Questionnaire | 6 months
  Impact on behavioural problems of women's other children will be assessed using the Strengths and Difficulties Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Van Lieshout, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- Strive Niagara, Welland, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No